CLINICAL TRIAL: NCT00968123
Title: Consecutive Series Outcomes Review of Patients Undergoing a New Single Portal Technique for Endoscopic Carpal Tunnel Release
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Charles Leinberry, MD, Rothman Institute
Other Study IDs: RIUCLEI 09-02
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Carpal Tunnel
MeSH Terms: conditions — Median Neuropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Purpose of this study is to report a new single portal endoscopic release technique and the sequence of the first 50 patients who underwent this release.

This will be a chart review of the demographics, outcomes, and complications of a sequential series of patients undergoing a Seg-Way Endoscopic carpal tunnel release (ECTR).

ELIGIBILITY:
Inclusion Criteria:

* This will be a chart review of the first 50 patients who have had surgery using the single portal technique

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This is a consecutive series, retrospective review of the first 50 patients who have undergone carpal tunnel release surgery using a new single portal endocopic technique.
Sampling Method: Probability Sample

PRIMARY OUTCOMES:
Functional outcomes following carpal tunnel release

SECONDARY OUTCOMES:
Complications and return to work data will also be reviewed

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States